CLINICAL TRIAL: NCT04923269
Title: A Single-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3532226 in Healthy Participants
Brief Title: A Study of LY3532226 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17834; J2V-MC-GZLA (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-06-09; First posted 2021-06-11 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12-15

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3532226 (Experimental): Single ascending doses of LY3532226 administered subcutaneously (SC).
  Interventions: Drug: LY3532226
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3532226 — Administered SC.
  Arms: LY3532226
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of the study drug known as LY3532226 in healthy participants. Blood tests will be performed to check how much LY3532226 gets into the bloodstream and how long it takes the body to eliminate it. This study will last approximately 8 weeks including screening period.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females not of childbearing potential.
* Body mass index (BMI) within the range of 18.5 to 40 kilograms per meter squared (kg/m²), inclusive

Exclusion Criteria:

* Have a significant history of or current CV (e.g., myocardial infarction, congestive heart failure, cerebrovascular accident, venous thromboembolism), respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk while taking the study intervention; or of interfering with the interpretation of data
* Have a history of malignancy within 5 years prior to screening
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis
* Have serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2X the upper limit of normal (ULN) or total bilirubin level (TBL) >1.5X ULN
* Have serum triglyceride level ≥5 mmol/L (442.5 mg/dL)
* Have undergone any form of bariatric surgery
* Have received systemic or inhaled glucocorticoid therapy (excluding topical, intraarticular, and intraocular preparations); for more than 14 consecutive days within 4 weeks before screening

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Week 8
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3532226 | Day 1 through Day 43
  PK: Cmax of LY3532226
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3532226 | Day 1 through Day 43
  PK: AUC of LY3532226
PK: Time to Maximum Concentration (Tmax) of LY3532226 | Day 1 through Day 43
  PK: Tmax of LY3532226

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No